CLINICAL TRIAL: NCT04066374
Title: Investigational Device Exemption for Intrathoracic Nerve Stimulation
Brief Title: Feasibility Study for Intrathoracic Nerve Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G190122
Record Dates: First submitted 2019-08-20; First posted 2019-08-26 (Actual); Results first posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-06

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment Arm (Experimental): Intrathoracic placement of neurostimulation device
  Interventions: Device: Peripheral Nerve Stimulation

INTERVENTIONS:
Device: Peripheral Nerve Stimulation — Medtronic Intellis Spinal Cord Stimulation Device to be implanted in thoracic cavity to treat postoperative acute pain.
  Other Names: Off-label use of Medtronic Intellis Spinal Cord Stimulation Device

SUMMARY:
The purpose of this study is to conduct an early clinical evaluation of safety and feasibility of peripheral nerve stimulation (PNS) of the intercostal nerves using an electrical lead placed in the thoracic cavity as a safe and effective method of pain control after cardiothoracic surgery.

DETAILED DESCRIPTION:
Despite minimally invasive techniques in thoracic surgery, postoperative pain can still be an issue for patients. Achieving adequate pain control not only affects a patient's short and long term quality of life but is also extremely important in preventing post-operative complications. Pain hinders with ambulating earlier and in performing pulmonary toilet hence increasing the risk of ensuing complications. While surgeons use multimodal approaches (e.g., epidural, regional anesthesia, NSAIDs, and opioids) to treat the postoperative pain, patients may not find relief in the acute period. Additionally, the use of opioids in the postoperative period can lead to chronic dependence and misuse. According to the Center for Disease Control, nearly 25% of patients chronically dependent on opioids started taking narcotics after they underwent a surgical procedure. Every day more than 115 people a day die from narcotics, and costing the United States $78.5 billion dollars a year. To prevent the need for opioids and their associated side effects, we look beyond medications for postoperative pain control.

The field of neuromodulation has been studying the effects of magnetic field and electrical current stimulation of different areas of the body to treat pain. While this has been shown to be effective for complex regional pain syndrome, low back pain, migraines and post herpetic neuralgia, there have not been studies applying the same concept to patients in the acute postoperative period. The goal is to apply the same concept of peripheral nerve stimulation to treat post thoracic surgery pain and decrease the need for opioids for pain relief.

The purpose of this investigational device exemption is to study the efficacy of peripheral nerve stimulation in treating post thoracic surgery pain and the safety of using these stimulation leads in the thoracic cavity.

ELIGIBILITY:
Inclusion Criteria:

• Patients undergoing pulmonary surgery by open thoracotomy or thoracoscopy with or without robotic assistance.

Exclusion Criteria:

* Woman who is pregnant,
* Subjects who have an active systemic infection or are immunocompromised,
* Subjects who will be exposed to diathermy or MRI,
* Subjects who have an electrically active implant, e.g., cardiac pacemaker, defibrillator, or neurostimulator,
* Subjects who are on anticoagulation therapy that would preclude their ability to undergo the implant procedure,
* Subjects less than 22 years of age,
* Subjects at elevated risk of infection or bleeding,
* Subjects unable to consent on their own,
* Subjects with active infection,
* Subjects with immunocompromised state,
* Subjects with preoperative chest pain,
* Subjects with pleural space infection or inflammatory process,
* Subjects undergoing esophageal, tracheal, or gastric procedures,
* Subjects undergoing pneumonectomy,
* Subjects with an uncorrectable coagulopathy,
* Subjects who are allergic or have shown hypersensitivity to any materials of the neurostimulation system which come in contact with the body.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sudish Murthy, MD PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Arm
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: years] | 65.8 [56 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 9
  Race: Other | 1
Baseline Pain Level [Mean (Full Range); unit: units on a scale] — Pain level expressed by the study subject in the scale of 0 (no pain) to 10 (unbearable pain). Lower scores represent the better outcome.
  units on a scale | 0 [0 to 0]

OUTCOME MEASURES:

1. Primary Outcome: Pain as Measured by the Visual-analog Scale
Description: Pain level expressed by the study subject in the scale of 0 (no pain) to 10 (unbearable pain). Lower scores represent the better outcome.
Time Frame: Baseline to 3 months
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 10
units on a scale | 1 [0 to 3]

2. Primary Outcome: Freedom From Device Related Adverse Events
Description: Freedom from device related adverse events (i.e., bleeding, infection, pneumothorax or arrhythmias)
Time Frame: up to 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 10
Participants
  Bleeding | 0
  Infection | 1
  Pneumothorax | 1
  Arrhythmias | 0

ADVERSE EVENTS:
Time Frame: Time of procedure to 3-months post-op visit
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=10)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=10)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Discomfort (General disorders) | 5 (5)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Discomfort (General disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/74/NCT04066374/Prot_SAP_000.pdf